CLINICAL TRIAL: NCT06670430
Title: Digital Heath Integration With Neuromodulation Therapies on Sensory and Motor Function in Patients With Diabetic Neuropathy
Brief Title: Digital Heath Integration With Neuromodulation Therapies on Diabetic Neuropathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Mohamed Abdelaty Marzouk, demonstrator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005260
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Diabetic Neuropathies
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Transcutaneous Electric Nerve Stimulation; Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): This group will include 30 type II diabetic patients with peripheral neuropathy Patients will receive TENS and NMES for 30 minutes 3 days per week,for 10 weeks with medical treatment
  Interventions: Device: experimental group
- control group (Placebo Comparator): This group will include 30 type II diabetic patients with peripheral neuropathy Patients will receive placebo TENS and NMES for 30-min sessions, 3 days per week, for 10 weeks with medical treatment
  Interventions: Device: control group

INTERVENTIONS:
Device: experimental group — This group will include 30 type II diabetic patients with peripheral neuropathy Patients will receive TENS and NMES for 30 minutes 3 days per week,for 10 weeks with medical treatment
  Other Names: TENS and NMES
  Arms: experimental group
Device: control group — This group will include 30 type II diabetic patients with peripheral neuropathy Patients will receive placebo TENS and NMES for 30-min sessions, 3 days per week, for 10 weeks with medical treatment
  Other Names: placebo TENS and NMES
  Arms: control group

SUMMARY:
This study will be carried out on 60 patients both gender male and female with diabetic neuropathy with age55-65 years. The patients will be selected from Elmahmoudia hospital .patients will be randomly assigned to two groups.

DETAILED DESCRIPTION:
Experimental Group:

This group will include 30 type II diabetic patients with peripheral neuropathy Patients will receive TENS and NMES for 30 minutes 3 days per week,for 10 weeks with medical treatment.

Control Group:

This group will include 30 type II diabetic patients with peripheral neuropathy Patients will receive placebo TENS and NMES for 30-min sessions, 3 days per week, for 10 weeks with medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Diagnosis of diabetes based on World Health Organization (WHO) with ages from 55to 65years 2. BMI> 25kg/m2 3. Clinically diagnosed with diabetic neuropathy. 4. All patients are taking oral hypoglycemic drugs with controlled diabetes mellitus.

  5. Willingness to comply with the study procedures and interventions. 6. Ability to provide informed consent. 7. presenting with Distal symmetric polyneuropathy (DSPN) based on a score of ≥7 on the validated Michigan Neuropathy Screening Instrument (MNSI) questionnaire.

  8. exhibiting moderately controlled blood pressure

Exclusion Criteria:

* 1. Presence of other significant neurological or musculoskeletal disorders that may confound the assessment of outcomes.

  2. Severe cognitive impairment or inability to provide informed consent. 3. Any recent surgical procedures or major medical events that could affect the study outcomes.

  4. Fracture. 5. Heart Failure. 6. Uncooperative patients. 7. Anemic patient. 8. Patients with liver diseases. 9. Smokers Patients. 10. Any cardiac pacemaker, automatic implantable cardioverter defibrillator (AICD), or other implanted electrical device 11. An existing deep vein thrombosis (DVT) 12. Any metal implants 13. Current foot ulceration or other lower limb skin ulcers 14. Any other cause of neuropathy

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-10 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
nerve conduction velocity | 10 weeks
  Adhesive patches called surface electrodes are placed on the skin over nerves or muscles at different spots. A very mild electrical impulse is applied via other patches or a handheld stimulator to stimulate the nerve.
  The resulting electrical activity of the nerve is recorded by the electrodes. The distance between electrodes and the time it takes for electrical impulses to travel between electrodes are used to measure the speed of the nerve signals. It is normal for several different nerves to be tested.
Electromyography | 10 weeks
  An EMG evaluates the electrical activity a muscle produces at rest and when it contracts, similar to an EKG of the heart muscle. The doctor places a single, small, Teflon-coated wire pin into selected muscles to be studied. The tip of the pin acts like an antenna, picking up electrical activity from the muscle that can be heard and seen on a screen. You will be asked to tighten (contract) the muscle. Electrical activity is recorded and can be heard as popping and clicking sounds when the muscle is contracting

SECONDARY OUTCOMES:
Google Fit | 10 weeks
  Google Fit is a mobile application developed by Google that focuses on tracking and monitoring physical activity and overall fitness. It is designed to help users lead healthier lifestyles by providing them with tools to set fitness goals, track their activity levels, and monitor their progress over time
Manage My Pain | 10 weeks
  Manage My Pain is a mobile application designed to assist individuals in tracking and managing chronic pain. It provides a comprehensive set of tools for users to monitor pain levels, treatments, and overall well-being. The app allows users to record detailed information about their pain, including intensity, location, triggers, and associated symptoms
PEDIS Score Diabetes App | 10 weeks
  PEDISScore is a mobile application developed for the assessment of diabetic neuropathy, a common complication of diabetes that affects the nerves. It is designed to assist healthcare professionals in evaluating the severity of diabetic neuropathy and monitoring its progression over time. The app utilizes the PEDISScore system

CONTACTS AND LOCATIONS:
Overall Officials: nesreen elnahas, phd, Study Chair — professor
Locations (1):
- Faculty of Physical Therapy, Dokki, Egypt